CLINICAL TRIAL: NCT03467685
Title: Determining the Variable Factors in Cutaneous Perception of Vibratory Stimulation
Brief Title: Variable Perception of Cutaneous Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Bryan Carroll, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Perception
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-08

CONDITIONS: Pain, Acute; Anesthesia, Local; Dermatology/Skin - Other
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned into one of two groups:
  Group 1: Vibratory anesthetic device (VAD) is in the OFF mode Group 2: VAD is in the ON mode
  We will use a random number generator to place patients into one of the two groups.
Who Masked: Participant
Masking Description: Subjects will be asked to close their eyes prior to the vibration anesthetic device (VAD) being applied to their skin. Only the user will know whether the VAD will be on or off based on the result of a random number generator. This will prevent anticipatory changes on the subjects side. The subject will be aware of the intervention after the device is turned on or left in the off position.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAD Off arm (Placebo Comparator): This will be the group that has the VAD placed on their skin in the off mode, i.e. no vibration
  Interventions: Device: Vibratory Anesthetic Device (VAD)
- VAD On arm (Experimental): This will be the group that has the VAD placed on their skin in the on mode, i.e. vibration
  Interventions: Device: Vibratory Anesthetic Device (VAD)

INTERVENTIONS:
Device: Vibratory Anesthetic Device (VAD) — This is a handheld ~10cm long tool, battery operated, which provides vibration at a rate of ~150 Hz

SUMMARY:
Perception of cutaneous sensory stimulation shows a large range of variability across multiple populations. Understanding this variability is critical to medical practice as interpretation of discomfort and pain is critical to diagnosis and treatment. Further, procedural medicine involves inflicting pain on patients in the form of injection of local anesthetic. Our protocol aims to determine how patients differentially interpret the non-noxious stimulation of vibration and the differences in perceiving anesthestic injection after the vibratory stimulus. We will explore how this ranges across all patients treated in a dermatological surgery out-patient setting. The goal is to identify which variables, such as age, gender, medical history, influence how sensation is interpreted.

ELIGIBILITY:
Inclusion Criteria:

* All patients

Exclusion Criteria:

* Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Falk Medical Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers. Data from this study may be used in future work.

REFERENCES:
- [Derived] Kazi R, Govas P, Slaugenhaupt RM, Carroll BT. Differential Analgesia From Vibratory Stimulation During Local Injection of Anesthetic: A Randomized Clinical Trial. Dermatol Surg. 2020 Oct;46(10):1286-1293. doi: 10.1097/DSS.0000000000002314. PMID 31895257
- [Derived] Govas P, Kazi R, Slaugenhaupt RM, Carroll BT. Effect of a Vibratory Anesthetic Device on Pain Anticipation and Subsequent Pain Perception Among Patients Undergoing Cutaneous Cancer Removal Surgery: A Randomized Clinical Trial. JAMA Facial Plast Surg. 2019 Dec 1;21(6):480-486. doi: 10.1001/jamafacial.2019.0733. PMID 31513234

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VAD Off Arm | VAD On Arm
Started | 52 | 49
Completed | 52 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAD Off Arm | VAD On Arm | Total
Number analyzed (Participants) | 52 | 49 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 28 | 52
  >=65 years | 28 | 21 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (1.1) | 66 (1.1) | 66 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 32 | 32 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 52 | 49 | 101
Location of treatment on body [Count of Participants; unit: Participants]
  Head and Neck | 38 | 34 | 72
  Trunk Extremities | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Score
Description: This is a tool used to measure the degree of pain perceived by the patient with application of the tool on their skin and following the injection of anesthetic which is part of the routine medical care of the patient. Score ranges from 0 to 10 with higher score indicating more pain.
Time Frame: Within 5 seconds of injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VAD Off Arm | VAD On Arm
Number analyzed (Participants) | 52 | 49
score on a scale | 2.0 (0.4) | 1.2 (0.2)
Statistical Analysis 1: Comparison: VAD Off Arm vs VAD On Arm; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Description: The definition of adverse events does not differ from that of clinicaltrials.gov.
Arm/Group | VAD Off Arm | VAD On Arm
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03467685/Prot_SAP_ICF_000.pdf